CLINICAL TRIAL: NCT01863589
Title: Drug Use Investigation for HEPSERA (Adefovir) Tablet
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112299
Record Dates: First submitted 2012-10-04; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — adefovir

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects prescribed adefovir tablets: Subjects with chronic hepatitis B or hepatic cirrhosis B to whom adefovir tablets are administered
  Interventions: Drug: Adefovir tablets

INTERVENTIONS:
Drug: Adefovir tablets — Administered according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
This post-marketing surveillance (PMS) is conducted to collect safety and efficacy data among subjects with chronic hepatitis B and hepatic cirrhosis B who is treated with adefovir tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic hepatitis B or hepatic cirrhosis B
* Subjects treated with adefovir tablets

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with chronic hepatitis B or hepatic cirrhosis B who are confirmed of hepatic function abnormality with continuous re-proliferation of hepatitis B virus while treated with lamivudine
Sampling Method: Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline